CLINICAL TRIAL: NCT02731196
Title: Comparison of Early Exercise Intervention Versus Late Exercise Intervention on Pain and Neurodynamic Mobility Following Unilateral Lumbar Microdiscectomy: A Randomized Controlled Trial
Brief Title: Comparison of Exercise Intervention Effects Following Lumbar Microdiscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Fahad AlKherayf, Neurosurgeon, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20150717-01H
Record Dates: First submitted 2016-04-01; First posted 2016-04-07 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Injury of Nerve Root of Lumbar and Sacral Spine
Keywords: exercise; lumbar microdiscectomy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early exercise intervention group (Experimental): Education, stabilization and neurodynamic level one exercises will be provided to the intervention group within one to two weeks following a unilateral lumbar microdiscectomy L3-4, L4-5, L5-S1. Within 4-6 weeks, this group will be provided with education, stabilization and neurodynamic level two exercises and a pedometer to monitor step count between week 4 and week 10 following the surgery.
  Interventions: Behavioral: Exercise Intervention
- Late exercise intervention group (Active Comparator): Education, stabilization and neurodynamic level one and two exercises will be provided to the active comparator group within 4-6 weeks following a unilateral lumbar microdiscectomy L3-4, L4-5, L5-S1. Within 4-6 weeks, this group will also be given instructions and a pedometer to monitor step count between week 4 and week 10 following the surgery.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Early versus later stabilization and neurodynamic exercise intervention following a post-op lumbar microdiscectomy

SUMMARY:
Low back pain is common, costly and affecting up to 80% of the population with the lumbar discectomy being a frequent spinal procedure for disc herniations. Pain & mobility impairments persist in patients following microdiscectomy with long term issues of back pain. The question remains as to why some patients recover quickly and without lasting difficulties while other patients persist with prolonged disability following the same surgery. The purpose of this study is to determine how to guide the patient towards full function and evaluate the timing to initiate strengthening, neurodynamics and a walking exercise program.

DETAILED DESCRIPTION:
The direction of treatment for low back pain both surgically and conservatively seeks to improve function in both daily and sporting activities for all patients. The patients continuing to suffer from a significant level of pain, disability and reduced function following single level microdiscectomy may benefit from a multi-factorial approach. A reduction in neurodynamic mobility related to dural adhesions is considered to be a contributing factor in this persistent peripheral neuropathic pain. The clinical efficacy of this study will address an exercise protocol post surgery in order to provide an optimal approach in the prevention of scar tissue that may be contributing to persistent pain post microdiscectomy. Mobility and motor control impairments are considered the consequence to the onset of pain. Education, neurodynamics and stabilization exercises are instrumental in the recovery post microdiscectomy with a reduction in pain and disability and the goal towards full functioning. The introduction of a neurodynamic protocol as an early exercise intervention may serve to reduce pain inhibition resulting with improved mobility and motor control. The recording of step count per day following a lumbar microdiscectomy will serve to document daily and physical activity levels following surgery. The purpose of this study is to determine whether or not there is a significant difference in pain levels and lumbar mobility between an early exercise intervention group versus a late exercise intervention group post microdiscectomy.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated unilateral post-op microdiscectomy L3-4, L4-5, L5-S1
* Radicular symptoms within one year of surgical intervention
* Ability to understand English or French for instructional purposes
* Able to participate in physical activity

Exclusion Criteria:

* Under the age of 18 years or over the age of 65 years
* Diagnosis of inflammatory conditions such as rheumatoid arthritis, ankylosing spondylitis
* Neoplasm
* Metabolic bone disease
* Cauda equine syndrome
* Neurological disorders ie Multiple Sclerosis, Parkinsons
* Compression of the spinal cord
* Uncontrolled cardiovascular or respiratory disease
* Peripheral vascular disease with sensory loss in the foot
* Discitis
* Pregnancy
* Previous spinal surgeries

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Oswestry Low Back Disability Questionnaire | 3 months
  Pain and function related to low back pain
Numeric Pain Rating Scale | 3 months
  Pain related to low back pain
Fear Avoidance Beliefs Questionnaire | 3 months
  Psychological barriers related to low back pain
Patient Specific Functional Scale | 3 months
  Function related to low back pain

SECONDARY OUTCOMES:
Lumbar mobility of flexion and extension | 3 months
  Range of lumbar motion related to low back pain
Slump test mobility | 3 months
  Mobility restrictions in the slump test related to low back pain
Straight leg raise | 3 months
  Mobility restrictions in the straight leg raise related to low back pain
50 ft Walk test | 3 months
  Time to complete 50 ft walk test
Step count per day | 4 weeks
  Step count per day related to Low back pain
Return to work | 3 months
  Timing for return to work related to low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alkherayf, MD MSc FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital - Civic Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Ottawa Hospital website — http://www.ottawahospital.on.ca